CLINICAL TRIAL: NCT03854591
Title: Gunshot Related Injuries in Trauma
Brief Title: A Snapshot Study of Patients Affected by Gunshot Related Injuries in Trauma in South Africa
Acronym: GRIT
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Dr Maritz Laubscher, Principal Investigator, University of Cape Town
Other Study IDs: 755/2018
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Trauma, Multiple; Gun Shot Wound
Keywords: GLOBAL SURGERY; COLLABORATIVE RESEARCH; GUNSHOT IN JURY; EPIDEMIOLOGY
MeSH Terms: conditions — Multiple Trauma; Wounds, Gunshot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gunshot related injury: Patients admitted to orthopaedic trauma service with gunshot related injury
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Introduction- Gun violence represents an important cause of disability to the working age population in South Africa. It has unrecognised, but undoubtedly significant implications for the health service and patients affected by these injuries.

Aim- To capture the burden of gunshot injury across South Africa and to establish a network of researchers in this field.

Method- A cross-sectional observational study run across South Africa capturing a nationwide picture of burden and complications associated with these injuries. Each centre will participate in a two-week window of patient screening and recruitment. Patients will be followed up at 6 weeks as per routine clinical practice. Data collected will include nature and number of treatments, length of stay, return to work and complications.

Results-Outcome of the study will be disseminated to the participating centres, relevant health boards and published with all contributors across centres recognised.

DETAILED DESCRIPTION:
Injury is a leading cause of death and morbidity in South Africa. It represents 8% of all cause mortality. Death by injury disproportionately affects young working age people who leave behind dependents. Those who survive their injury may suffer long standing disability. However funding for research in injury accounts for less than 1% percent of the research expenditure of the MRC South Africa. This is particularly incongruous as 'injury' was identified by the Essential National Health Research congress as the number 1 priority for the MRC as far back as 1996.

Causes of injury include work related injury, road accidents and interpersonal violence. Within interpersonal violence, gunshot injuries are a particularly lethal and disabling. South Africa has the 18th highest number of gun owners in the world. However it has a gun homicide rate of 8.2 per hundred thousand. This is comparable to the United States, which has the highest levels of gun ownership anywhere in the world.

This is also the highest number anywhere in Southern Africa. It places South Africa amongst some of the most violent countries in the world such as Honduras and Brazil.

The legacy of gun injuries can be just as devastating to communities with persistent disability and escalating feuds. The health impact of gun related injury has been explored in a few specific centres however the broader national picture remains unclear (4). It seems likely that specific areas will bear most of the gun problem. If this can be sufficiently understood specific interventions resources and expertise can be most appropriately deployed.

RATIONALE FOR CURRENT STUDY Gunshot related injuries are an important cause of mortality and morbidity. In South Africa, this burden is under studied and relatively unique. Most studies focus on death as an outcome for gun related violence, however injuries to limbs as seen by orthopaedic teams are rarely fatal. Unfortunately such injuries are highly significant and cause long term disability for patients. Gunshot injuries are also very resource intensive to treat.

Injury is a significant research priority for South Africa, but currently it receives little funding. There are also no structures in place to study injury and its treatment on a nationwide basis.

This study seeks to build such a network around the clinical problem of gunshot injury. In turn this will act as a platform to deliver big and important clinical effectiveness research for future generations of South African patients.

STUDY OBJECTIVES Primary- To capture on a nationwide basis the burden of orthopaedic gunshot injury in patients.

Secondary- To establish a research collaborative network for Orthopaedic trauma across South Africa.

STUDY METHOD A snap shot cohort study run across participating sites in South Africa. All sites in South Africa offering orthopaedic care have been invited to participate. Each will return anonymised routine data on patients who meet the eligibility criteria over a two week study window. Each patient will be approached for consent as detailed below.

Once open each site will be responsible for recording each patient that meets the inclusion criteria that is referred to the trauma and orthopaedic service.

Outcomes collected will aim to inform both patient level and healthcare system costs in terms of burden of work and legacy of injury.

Each patient will have a unique alphanumeric study number. Against this anonymous identifier, the site data collector(s) will record the data on a secure web based database (REDCap). This safe and secure method will return data to the study coordinating centre.

Consent Each patient will be approached and consent to participate sought. This will cover their agreement to have data recorded; to answer additional questions related to the research objectives both at admission and at follow up. Consent forms will be stored locally. Where patients lack capacity to consent on admission, they will be recorded on the study screening log anonymously. For the duration of their inpatient stay, the clinical team will assess them for recovery of capacity. If the patient dies or fails to recover then only the anonymous screening log data will be recorded in the study. A final attempt to recruit the patient will be made at the 6 week follow up appointment.

ELIGIBILITY:
Inclusion Criteria:

* Any gunshot related injury presenting to registered study hospital's orthopaedic service.

Exclusion Criteria:

* Isolated injuries to the head, chest or abdomen
* Patients under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any adult patient presenting with at least one gunshot injury to the limb, spine or pelvis
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Destination at discharge | 6 weeks after enrolment to study date
  Record of alive, dead or discharged

SECONDARY OUTCOMES:
Number of cases | 18/02/2019-04/03/2019
  Total number of gunshot related injuries admitted at each unit
Return to follow up | 01/04/2019-15/04/2019
  Number of patients that attend their routine follow up appointment
Number of patients who give consent to additional study questions | 18/02/2019-04/03/2019
  Each patient with capacity will be asked to give consent to ask additional questions
Health Related Quality of Life | Total study period 18/02/2019-15/04/2019
  Baseline and follow up HRQOL will be assessed using the EQ5D assessment where patients have given consent
Complications | Total study period 18/02/2019-15/04/2019
  At 6-8 week after index admission window any noted complications will be recorded (including surgical site infection and failure of fixation)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Graham, FRCS, Principal Investigator — Liverpool School of Hygiene and Tropical Medicine; Sithombo Maqungo, FCS, Principal Investigator — UCT; Michael Held, FCS, Principal Investigator — UCT; Maritz Laubscher, FCS, Principal Investigator — UCT; James Masters, MRCS, Principal Investigator — University of Oxford
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa